CLINICAL TRIAL: NCT06547827
Title: Rehabilitation With and Without Robot and Allied Digital Technologies (RADTs) in Stroke Patients: a Pragmatic Multicenter Randomised Controlled Trial on the Effectiveness, Acceptability, Usability, and Economic-organizational Sustainability of RADTs From Subacute to Chronic Phase
Brief Title: Rehabilitation With and Without Robot and Allied Digital Technologies in Stroke Patients
Acronym: StrokeFit4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Istituti Clinici Scientifici Maugeri SpA (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Ospedale Policlinico San Martino (Other); Università di Pavia (Unknown); Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIT4MedRobStroke; PNC0000007 (Other Grant/Funding Number: Ministry of University and Research of Italy)
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: rehabilitation; robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Treatment with Robotic & Technological Devices (RADTs) (Experimental): This intervention employs various RADTs to target the following domains: a) upper limb sensorimotor abilities; b) lower limb sensorimotor abilities and gait; c) balance; and d) cognitive abilities. For upper limb sensorimotor function, we will use planar end-effector robots, exoskeletons, or electromechanical systems for shoulder, elbow, and wrist rehabilitation; end-effector robots or exoskeletons for hand rehabilitation; and sensor-based devices for comprehensive upper limb treatment. For lower limb sensorimotor function, we will utilize end-effector robots or exoskeletons and treadmills with body-weight support systems. Balance training will involve stabilometric platforms and sensor-based systems. Cognitive functions will be addressed using digital systems, sensor-based devices, and virtual reality programs. All devices must have a CE mark for medical devices and be used according to the manufacturer's specifications.
  Interventions: Other: robotic rehabilitation
- Traditional Treatment (Active Comparator): In the control group, subjects will undergo a standard traditional rehabilitation program without the use of RADTs, focusing on the following domains:a) upper limb sensorimotor abilities; b) lower limb sensorimotor abilities and gait; c) balance; and d) cognitive abilities, using traditional methods of physiotherapy and cognitive rehabilitation.
  Interventions: Other: traditional rehabilitation

INTERVENTIONS:
Other: robotic rehabilitation — Treatment will occur in a gym equipped with devices for all the domains, with two physiotherapists supervising groups of 4 to 6 patients, depending on their clinical severity.
  Patients will undergo a total of 25 sessions, each lasting 45 minutes, with the following frequency:
  * 5 times a week for 5 weeks, for inpatients;
  * 3 times a week for 8.3 weeks, for outpatients.
  Arms: Integrated Treatment with Robotic & Technological Devices (RADTs)
Other: traditional rehabilitation — A physiotherapist-to-patient ratio of 1:1 is provided for the treatment in all participating centres.
  Patients will undergo a total of 25 sessions, each lasting 45 minutes, with the following frequency:
  * 5 times a week for 5 weeks, for inpatients;
  * 3 times a week for 8.3 weeks, for outpatients.
  Arms: Traditional Treatment

SUMMARY:
Rehabilitation after stroke often employs Robot and Allied Digital Technologies (RADTs), yet evidence on their effectiveness remains inconclusive due to study heterogeneity and limited sample sizes.

This multicentre randomized controlled pragmatic trial aims at comprehensively and accurately assessing the effectiveness of rehabilitation mediated by RADTs after a stroke, compared to traditional rehabilitation, also considering economic sustainability.

DETAILED DESCRIPTION:
The aim of this study is to evaluate, in a pragmatic trial on a large sample of patients who have experienced a stroke within the six months prior to enrollment, the effectiveness of a multimodal treatment using robotics and advanced technologies compared to traditional multimodal treatment, in the recovery of activities of daily living.

Primary Objective: To demonstrate, in a population of subacute stroke patients, the non-inferiority of a rehabilitation treatment integrated with robotic and/or technological devices compared to traditional rehabilitative treatment in the recovery of activities of daily living.

Secondary Objectives:

* To demonstrate the superiority of rehabilitative treatment integrated with robotic and/or technological devices compared to traditional rehabilitation treatment in the recovery of activities of daily living, should non-inferiority be demonstrated;
* To compare the improvements between two groups in all targeted domains (upper limb sensorimotor abilities; lower limb sensorimotor abilities and gait; balance; cognitive abilities), in accordance with the International Classification of Functioning, Disability, and Health (ICF);
* To analyze the neurophysiological parameters and factors involved in neuroplasticity processes;
* To compare the time pattern of manual dexterity and walking performance recovery in the two groups;
* To assess the effects of the rehabilitation treatment in terms of daily life activities and quality of life through medium-term follow-up;
* To evaluate the acceptability and usability of the rehabilitative treatment integrated with robotic and/or technological devices for the patient, their family, and the healthcare practitioner;
* To create a predictive model capable of forecasting the effectiveness of robotic and technological treatment in subjects after a stroke, based on a detailed description of the patient at baseline (using demographic data and clinical picture at admission);
* To assess the economic sustainability of the rehabilitative treatment integrated with robotic and/or technological devices for the patient, payer, and society, through the creation of a model for the assessment and prediction of cost-effectiveness, cost-utility, and, for the healthcare system, a Budget Impact Analysis, and related sensitivity analyses.

The study employs a multicenter, multimodal, randomized, controlled, parallel-group (1:1) interventional design with blinded assessors, following a pragmatic approach. It will be conducted across multiple clinical centers involved in a national research initiative, encompassing both outpatient and inpatient settings. Randomization will be centralized and stratified by clinical center, latency, and clinical setting (inpatients or outpatients).

The sample size (596 patients) was determined considering the following, with respect to the primary outcome (the change in the modified Barthel Index): (a) the non-inferiority of robotic treatment compared to traditional treatment; (b) a power of 80%; (c) a non-inferiority margin of 5 points; (d) a bilateral 95% confidence interval; (e) a standard deviation of the primary outcome of 20 points. Considering these parameters, a sample size of 506 patients (253 per group) is obtained. Additionally, considering a dropout rate of 15%, a total sample size of 596 patients is obtained. The same sample size is sufficient to also demonstrate the potential superiority of robotic treatment. In fact, considering a significance level of 5%, a power of 80%, a minimal clinically important difference of the scale of 9.25 points, a standard deviation of 20 points, and a dropout rate of 15%, a total of 178 patients are required for demonstrating superiority.

The experimental group will receive rehabilitation using RADTs within a new organizational model, where two physical therapists supervise four to six patients. In the control group, patients will undergo individual traditional rehabilitation, maintaining a 1:1 patient-to-therapist ratio. In both groups, patients will undergo comprehensive rehabilitation treatment, targeting the following domains: a) upper limb sensorimotor abilities; b) lower limb sensorimotor abilities and gait; c) balance; d) cognitive abilities.

The primary outcome is to demonstrate non-inferiority in activities of daily living as measured by the modified Barthel Index. Should non-inferiority be established, the study will then evaluate the potential superiority of RADTs in activities of daily living.

All participating centers will follow a standardized operating procedure regarding treatment and outcome assessment to ensure consistency across all sites. Data will be systematically collected using the REDCap (Research Electronic Data Capture) platform.

ELIGIBILITY:
Inclusion Criteria:

* First-ever diagnosis of ischemic or haemorrhagic stroke confirmed by Computed Tomography or Magnetic Resonance Imaging;
* Age 18 years and over;
* Time since the event equal to or less than 6 months;
* Mild to severe impairment of the upper limb (motor section of the Fugl-Meyer Assessment of Upper Extremity ≤ 58) and/or mild to severe impairment of the lower limb (score on the Functional Ambulation Categories scale ≤ 4) and/or mild to severe impairment of balance (Berg Balance Scale ≤ 45);
* Clinical stability allowing transfer to the gym and execution of the planned treatments.

Exclusion Criteria:

* Clinical instability;
* Behavioral/cognitive disorders preventing adequate patient compliance with both traditional and robotic rehabilitation treatment (severe cognitive deficit, Montreal Cognitive Assessment <10);
* Rigidity or hypertonia (Modified Ashworth Scale > 3) in the plegic/paretic limb;
* Serious uncorrectable visual impairments preventing the patient from performing treatment with technological and/or robotic devices;
* Pregnant women;
* Refusal to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the modified Barthel Index | baseline; within 24 hours from the 25th rehabilitation session
  The modified Barthel Index for Activities of Daily Living is a validated ordinal scale which measures a person's ability to complete activities of daily living (ADL). Scores range from 0 (total dependence) to 100 (total independence).

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for the upper extremities - motor function | baseline; within 24 hours from the 25th rehabilitation session
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The upper extremity motor function domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist, and hand. It ranges from 0 (hemiplegia) to 66 (normal motor performance).
Fugl-Meyer Assessment for the upper extremities - sensory function | baseline; within 24 hours from the 25th rehabilitation session
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The upper extremity sensory function domain evaluates light touch on two surfaces of the arm, and position sense for upper limb joints. It ranges from 0 to 12 (normal sensory function).
Fugl-Meyer Assessment for the lower extremities - motor function | baseline; within 24 hours from the 25th rehabilitation session
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The lower extremity motor function domain includes items assessing movement, coordination, and reflex action of the hip, knee, and ankle. It ranges from 0 (hemiplegia) to 34 (normal motor performance).
Fugl-Meyer Assessment for the lower extremities - sensory function | baseline; within 24 hours from the 25th rehabilitation session
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The lower extremity sensory function domain evaluates light touch on two surfaces of the leg, and position sense for lower limb joints. It ranges from 0 to 12 (normal sensory function).
Berg Balance Scale | baseline; within 24 hours from the 25th rehabilitation session
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14-item scale designed to measure balance of the older adult in a clinical setting. It ranges from 0 to 56. A higher score indicates better balance.
Symbol Digit Modalities Test | baseline; within 24 hours from the 25th rehabilitation session
  The Symbol Digit Modalities Test evaluates information processing speed. It consists of a simple task of replacing symbols with numbers. Using a reference key, the patient has 90 seconds to match a sequence of symbols with the correspondent numbers as rapidly as possible. Both written or oral administration can be used. For each correct answer, a point is assigned. The higher the score, the faster the information processing speed.
Modified Ashworth Scale | baseline; within 24 hours from the 25th rehabilitation session
  The Modified Ashworth Scale (MAS) is a revised version of the original Ashworth Scale that measures spasticity in patients with lesions to the central nervous system. MAS is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0 to 4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch. The lower the score, the lower the spasticity. Upper and lower joints spasticity is assessed.
Motricity Index for upper extremities | baseline; within 24 hours from the 25th rehabilitation session
  The Motricity Index (MI) is an ordinal method of measuring limb strength. For upper extremity test, shoulder abduction, elbow flexion, pinch grip are considered. It ranges from 0 (worse) to 100 (normal strength).
Motricity Index for lower extremities | baseline; within 24 hours from the 25th rehabilitation session
  The Motricity Index (MI) is an ordinal method of measuring limb strength. For lower extremity test, hip flexion, knee extension, and ankle dorsiflexion are considered. It ranges from 0 (worse) to 100 (normal strength).
Trunk control test | baseline; within 24 hours from the 25th rehabilitation session
  The Trunk control test (TCT) measures four simple aspects of trunk movement. Total score range from 0 (minimum) to 100 (maximum, indicating better performance).
Numerical Rating Scale for Pain | baseline; within 24 hours from the 25th rehabilitation session
  The Numerical Rating Scale fo Pain (NRSP) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Neuropathic Pain 4 Questions | baseline; within 24 hours from the 25th rehabilitation session
  The Neuropathic Pain 4 Questions (DN4) is a validated clinician-administered screening tool for neuropathic pain. It ranges from 0 to 10; higher values means higher neuropathic pain probability.
Action Research Arm test | baseline; within 24 hours from the 25th rehabilitation session
  The Action Research Arm Test (ARAT) is a 19 item observational measure used to assess upper extremity performance (coordination, dexterity and functioning). The 19 items comprising the ARAT are scored using a 4 point ordinal scale. Scores on the ARAT may range from 0-57 points, with a maximum score of 57 points indicating better performance.
2 Minute Walk Test | baseline; within 24 hours from the 25th rehabilitation session
  The 2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity. The person is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured.
5-level EQ-5D | baseline; within 24 hours from the 25th rehabilitation session
  The 5-level EQ-5D (EQ-5D-5L) is a validated tool to assess health-related quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Index scores range from -0.59 to 1; 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.
Brain Symmetry Index | baseline; within 24 hours from the 25th rehabilitation session
  The Brain Symmetry Index (BSI) is a quantitative electroencephalographic (qEEG) measure used to assess the degree of symmetry in brain activity between the two hemispheres. It is defined as the mean absolute difference in spectral power of the EEG signals from homologous channels pairs on the left and right hemispheres, in the frequency range from 1 to 25 Hz. A higher BSI value indicates greater asymmetry, which is often associated with poorer clinical outcomes in stroke patients.
Delta/Alpha Ratio | baseline; within 24 hours from the 25th rehabilitation session
  The Delta/Alpha Ratio (DAR) is a quantitative electroencephalographic (qEEG) measure used to assess the balance between slow-wave (delta) and fast-wave (alpha) brain activity. It is calculated by dividing the power of delta waves (0.5-4 Hz) by the power of alpha waves (8-12 Hz). The DAR is particularly useful in evaluating brain function in stroke patients, as an increased DAR is often associated with greater brain dysfunction and poorer clinical outcomes.
Change in serum concentration of Glial Fibrillary Acidic Protein (GFAP) | baseline; within 24 hours from the 25th rehabilitation session
  Serum GFAP Concentration will be evaluated by "Ella" automated Immunoassay System method.
Serum concentration of Neurofilament light (NfL) | baseline; within 24 hours from the 25th rehabilitation session
  Serum NfL Concentration will be evaluated by "Ella" automated Immunoassay System method.
Serum concentration of Brain Derived Neurotrophic Factor (BDNF) | baseline; within 24 hours from the 25th rehabilitation session
  Serum BDNF Concentration will be evaluated by "Ella" automated Immunoassay System method.
10 Meter Walk Test | baseline; within 24 hours from: the 5th rehabilitation session; the 10th rehabilitation session; the 15th rehabilitation session; the 20th rehabilitation session; the 25th rehabilitation session
  The 10 Meter Walk Test is a performance measure used to assess walking or gait speed in meters per second over a distance of 10 meters
Box and block test | baseline; within 24 hours from: the 5th rehabilitation session; the 10th rehabilitation session; the 15th rehabilitation session; the 20th rehabilitation session; the 25th rehabilitation session
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. The individual is instructed to move as many blocks as possible, one at a time, from one compartment to the other of a test box with 150 blocks and a partition in the middle. The number of blocks transferred in 60 seconds is recorded. Both the affected and the not affected side are measured.
modified Barthel Index (follow-up) | 1 month after the end of the treatment; 2 months after the end of the treatment; 3 months after the end of the treatment; 4 months after the end of the treatment; 5 months after the end of the treatment; 6 months after the end of the treatment;
  The Barthel Index for Activities of Daily Living is a validated ordinal scale which measures a person's ability to complete activities of daily living (ADL). Scores range from 0 (total dependence) to 100 (total independence).
EQ-5D-5L (follow-up) | 1 month after the end of the treatment; 2 months after the end of the treatment; 3 months after the end of the treatment; 4 months after the end of the treatment; 5 months after the end of the treatment; 6 months after the end of the treatment;
  The 5-level EQ-5D version (EQ-5D-5L) is a validated tool to assess health-related quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Index scores range from -0.59 to 1; 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.

OTHER OUTCOMES:
premorbid Modified Rankin Scale | At baseline
  The pre-stroke Modified Rankin Score (mRS) is an estimated score used to assess the patient's pre-stroke level of function. It has a grade ranging from 0 (no symptoms) to 6 (dead).
Life Time Physical Activity Questionnaire | At baseline
  The Life Time Physical Activity Questionnaire (LTPAQ) is an interviewer-administered questionnaire used to estimate a respondent's physical activity done from childhood to the present.
Cognitive Reserve Index | At baseline
  The Cognitive Reserve Index questionnaire (CRIq) aims to collect and estimate the amount of cognitive reserve acquired during a person's lifetime. In a single index (CRI), the questionnaire conveys three main sources of cognitive reserve: education, working activity, and leisure time activities. The CRIq score fell into 1 of 5 ordered levels: low (less than 70); medium-low (70-84); medium (85-114); medium-high (115-130); and high (more than 130).
National Institutes of Health Stroke Scale (NIHSS) | At baseline
  It is validated tool for assessing stroke severity. NIHSS scores range from 0 to 42, with higher scores indicating more severe neurological deficit.
Cumulative Illness Rating Scale - severity index | At baseline
  The Cumulative Illness Rating Scale (CIRS) is a well-validated multidimensional test commonly used as part of the Comprehensive Geriatric Assessment. It offers a comprehensive disease assessment for 14 organ systems, based on a rating scale ranging from 0 (best) to 4 (worst) for each. The severity index (CIRS-SI) is the mean of the scores of the first 13 categories (excluding the category of psychiatric/behavioral pathologies), ranging then from 0 to 4.
Cumulative Illness Rating Scale - comorbidity index | At baseline
  The Cumulative Illness Rating Scale (CIRS) is a well-validated multidimensional test commonly used as part of the Comprehensive Geriatric Assessment. It offers a comprehensive disease assessment for 14 organ systems, based on a rating scale ranging from 0 (best) to 4 (worst) for each. The comorbidity index (CIRS-CI) is the number of categories in which a score greater than or equal to 3 is obtained (excluding the category of psychiatric/behavioral pathologies). This index ranges from 0 to 13, with 0 indicating no significant comorbidity and 13 indicating severe comorbidity in all categories.
Thumb Localizing Test | At baseline
  It is a standardised measure of proprioception. It ranges from 0 (normal) to 3.
Semmes Weinstein filament test | At baseline
  It measure the level of light touch sensation of the tips of the thumb and index finger. The Semmes Weinstein filament test kit consists of 20 flexible nylon monofilaments of constant length, but varying in diameter. They are labeled so as to give a linear scale of perceived intensity (1.65-6.65) using a logarithmic scale of applied force: labeled number = Log10 of (10 × force in milligrams). The more the labeled number increases, the thicker the filament becomes, and the more pressure is necessary to bend the filament, meaning lower level of light touch sensation.
Fatigue Severity Scale | At baseline
  The Fatigue Severity Scale(FSS) is a nine-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. The scale addresses fatigue's effects on daily functioning, querying its relationship to motivation, physical activity, work, family, and social life, and asking respondents to rate the ease with which they are fatigued and the degree to which the symptom poses a problem for them. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score is 9 and maximum score possible is 63. Higher score indicate greater fatigue severity.
Blaylock Risk Assessment Screening Score | At baseline
  It is a simple and easy to use instrument that explores some important risk factors, such as social support, functional status, number of active medical problems and number of drugs, to identify the risk of prolonged hospitalization and the need of discharge planning in individuals who are hospitalized. It comprises a 10-item scale that determines a score between 0 and 40: a result lower than 10 identifies patients which have few needs for discharge planning and a low demand for discharge planning resources.
Montreal Cognitive Scale | At baseline
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. It ranges from 0 (worst) to 30 (best).
Intrinsic Motivation Inventory | within 24 hours from the 5th rehabilitation session
  The Intrinsic Motivation Inventory (IMI) is a questionnaire that provides qualitative information on the content and level of motivation that an user experiences during an intervention Each IMI item consists of a seven-point Likert scale, ranging from "not at all true" to "completely true", with a maximum score of 144. Higher scores mean a more positive result on motivation.
Hospital Anxiety and Depression Scale | At baseline
  It is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic. The Hospital Anxiety and Depression Scale (HADS) is a 14-question instrument that measures anxiety and depression. Each question is scored between 0 (no impairment) and 3 (severe impairment), with a maximum score of 21 for anxiety or depression.
Beck Depression Inventory | At baseline
  The Beck Depression Inventory (BDI-II), is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. The range of possible scores is 0 to 63. BDI-II scores are classified as minimal (0-13), mild (14-19), moderate (20-28), and severe (29-63) depression.
Mini Nutritional Assessment Short-Form | At baseline
  It is a validated questionnaire for nutritional assessment. The total score range from 0 to 14 points, with scores of 12 to 14 points indicating normal nutritional status, scores between 8 and 11 points identifying patients at risk of malnutrition, and scores < 8 points diagnosing malnutrition.
SARC-F | At baseline
  The SARC-F questionnaire is a screening tool to identify probable sarcopenic patients. The questionnaire screens patients for self-reported signs suggestive of sarcopenia, which include deficiencies in strength, walking, rising from a chair, climbing stairs, and experiencing falls. Each of the self-reported parameters receives a minimum and maximum score of 0 and 2, respectively, with the greatest maximum SARC-F score being 10.
Functional Oral Intake Scale | At baseline
  It is a tool to assess functional oral intake of food and liquids in patients with oropharyngeal dysphagia.specifically, it is a 7-point ordinal scale describing the functional level of oral intake of food and liquids. Level 7 represents a full oral diet with no restrictions, levels 6-4 indicate a full oral diet with restrictions, levels 3-2 describe a mixed oral and tube intake, while level 1 represents a totally tube-dependent intake.
Handgrip test | At baseline
  It is an instrumented measure of grip strength.
Number of patients with the Brain Derived Neurotrophic Factor (BDNF) genetic polymorphism rs6265 (Val66Met) classified by genotype: homozygous GG (Valine/Valine), heterozygous GA (Valine/Methionine), or homozygous AA (Methionine/Methionine). | At baseline
  It is a genetic analysis of BDNF polymorphism rs6265; it is performed using the HpyCH4IV restriction enzyme on DNA extracted from whole blood and amplified with PCR reaction. The polymorphism rs6265 identifies homozygous Valine/Valine, heterozygous Valine/Methionine and homozygous Methionine/Methionine.
5-level EQ-5D | baseline; within 24 hours from the 15th rehabilitation session; within 24 hours from the 25th rehabilitation session
  The 5-level EQ-5D (EQ-5D-5L) is a validated tool to assess health-related quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Index scores range from -0.59 to 1; 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.
Computer skills questionnaire | At baseline
  It is an ad-hoc questionnaire to assess computer skills.
Technology Acceptance Model | within 24 hours from the 5th rehabilitation session; within 24 hours from the 15th rehabilitation session; within 24 hours from the 25th rehabilitation session
  It is a questionnaire used with the primary aim of identifying the determinants involved in the acceptance of Robotic and Allied Technology. The questionnaire consists of 4 sections (perceived usefulness, ease of use, compatibility, intention to use); each question includes a 7-point Likert scale, from 1 (worst) to 7 (best). The scoring is calculated for each section and is given by the average of the responses in that section, ranging from 1 (worst) to 7 (best).
Questionnaire for satisfaction | baseline; within 24 hours from the 25th rehabilitation session
  This is an ad-hoc questionnaire designed to measure satisfaction with healthcare services. Each question uses a 5-point Likert scale, ranging from 1 (unsatisfied) to 5 (very satisfied).
Questionnaire for perception of problems and solution complexity | baseline; within 24 hours from the 25th rehabilitation session
  It is an ad-hoc questionnaire for perception of problems and solution complexity. Each question utilizes a 5-point Likert scale, ranging from 1 (low complexity) to 5 (very complex).
Questionnaire for costs | baseline; within 24 hours from the 15th rehabilitation session; within 24 hours from the 25th rehabilitation session
  Ad-hoc questionnaire to evaluate the costs (direct healthcare costs, direct non-healthcare costs, indirect costs ) incurred by the patient.
Incremental cost-utility ratio | During the study,an average of 24 months
  The incremental cost-utility ratio (ICUR) will serve as the key metric of the Cost-utility analysis, and it is calculated as the ratio between differences in costs and differences in utility across the analysis groups. Cost-utility analysis will assess and compare the efficiency of alternative rehabilitation interventions by measuring health outcomes in terms of utility, a measure of general well-being or quality of life (subjective measures), relative to the costs incurred to achieve these outcomes. Utilities will be evaluated using standardized measures based on quality of life. Each health condition identified through generic health-related quality of life questionnaires (EQ-5D-DL) will be associated with available utility scores specific to Italy.
Incremental cost-effectiveness ratio | During the study, an average of 24 months
  The incremental cost-effectiveness ratio (ICER) is calculated by dividing the difference in costs between the alternative rehabilitation models tested in the clinical study by the difference in clinical outcomes (physical units - objective measures). It will be used as the key metric of the cost-effectiveness analysis, that will compare the costs and clinical outcomes of the alternative rehabilitation models being studied. The ICER represents the additional cost incurred to achieve an incremental unit of effectiveness, that will be assessed considering primary and secondary outcomes.
Financial impact (differences in direct health costs) | During the study, an average of 24 months
  From the perspective of the payer, the expected outcome of the budget impact analysis is the assessment of the financial impact (differences in direct health costs) over a 3-5 year period for the diffusion of a mix of robotic-based rehabilitations, compared to conventional rehabilitation or a robotic solution. The financial impact will be assessed by considering the direct health costs associated with the different rehabilitation regimes, varying projections of robotic market uptake, and the degrees of substitutability between the compared rehabilitation regimes.

CONTACTS AND LOCATIONS:
Overall Officials: Irene G Aprile, Study Director — IRCCS Fondazione Don Carlo Gnocchi; Irene G Aprile, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi; Christian Lunetta, Principal Investigator — IRCCS Istituti Clinici Scientifici Maugeri; Roberto De Icco, Principal Investigator — IRCCS Fondazione Mondino; Carlo Trompetto, Principal Investigator — IRCCS Ospedale Policlinico San Martino; Silvana Quaglini, Principal Investigator — Università di Pavia; Giuseppe Turchetti, Principal Investigator — Scuola Superiore Sant'Anna di Pisa
Locations (13):
- Italy (13):
  - Fondazione Don Carlo Gnocchi, Centro Gala, Acerenza
  - IRCCS Istituti Clinici Scientifici Maugeri, Bari
  - IRCCS Ospedale Policlinico San Martino,, Genova
  - Fondazione Don Carlo Gnocchi, IRCCS Santa Maria Nascente, Milan
  - IRCCS Istituti Clinici Scientifici Maugeri, Milan
  - IRCCS Istituti Clinici Scientifici Maugeri, Montescano
  - IRCCS Fondazione Mondino, Pavia
  - IRCCS Istituti Clinici Scientifici Maugeri, Pavia
  - Fondazione Don Carlo Gnocchi, Centro Santa Maria della Provvidenza, Roma
  - Fondazione Don Carlo Gnocchi, Centro Santa Maria al Mare, Salerno
  - Fondazione Don Carlo Gnocchi, Polo Specialistico Riabilitativo, Sant'Angelo dei Lombardi
  - IRCCS Istituti Clinici Scientifici Maugeri, Telese Terme
  - Fondazione Don Carlo Gnocchi, Polo specialistico riabilitativo, Tricarico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the publication will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning six months after the publication, with no end date.
Access Criteria: Access will be provided to the general scientific community and any interested researchers, for any type of analysis or secondary research use. The data will be made available on a public data-sharing platform such as Zenodo, or Figshare.

REFERENCES:
- [Derived] Aprile IG, Germanotta M, Fasano A, Siotto M, Mauro MC, Pavan A, Nicora G, Sgandurra G, Malovini A, Oreni L, Dubbini N, Parimbelli E, Comande G, Lunetta C, Fiore P, De Icco R, Trompetto C, Trieste L, Turchetti G, Quaglini S, Messa C; STROKEFIT4 Study Group. Rehabilitation with and Without Robot and Allied Digital Technologies (RADTs) in Stroke Patients: A Study Protocol for a Multicentre Randomised Controlled Trial on the Effectiveness, Acceptability, Usability, and Economic-Organisational Sustainability of RADTs from Subacute to Chronic Phase (STROKEFIT4). J Clin Med. 2025 Apr 15;14(8):2692. doi: 10.3390/jcm14082692. PMID 40283522